CLINICAL TRIAL: NCT01586299
Title: The Role of Non Steroidal Anti Inflammatory Drugs in the Treatment of Pleuropneumonia in Children. a Randomized Controlled Trial
Brief Title: NSAIDs Treatment in Children With Pleuropneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 262-11-RMC
Record Dates: First submitted 2012-03-19; First posted 2012-04-26 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2012-01

CONDITIONS: Pleuro-pneumonia
Keywords: pleuropneumonia children; non steroidal anti inflammatory drugs; pleural effusion; severe pneumonia
MeSH Terms: conditions — Pleural Effusion; Pneumonia | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ibuprofen (Experimental)
  Interventions: Drug: Ibuprofen
- acetaminophen (Active Comparator)
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — 10 mg/kg every 8 hours until 24 hours after resolution of fever
  Other Names: nurofen; advil
  Arms: ibuprofen
Drug: Acetaminophen — 15 mg/kg every 6 hours until 24 hours after resolution of fever
  Other Names: paracetamol; acamol
  Arms: acetaminophen

SUMMARY:
The purpose of this study is to evaluate the influence of routine NSAIDs treatment for hospitalized children with pleuropneumonia in comparison with acetominophen treatment (all in conjunction with adequate antibiotic therapy).

ELIGIBILITY:
Inclusion Criteria:

* age less than 18 years
* admission in Schneider childrenMC of Israel, wards a/c
* clinical diagnosis of pneumonia with evidence of pleural effusion on chest X-ray
* parental informed consent
* follow-up ability after discharge

Exclusion Criteria:

* pneumonia secondary to foreign body aspiration
* immune deficiency
* chronic lung disease other than asthma (CF, CLD of prematurity, Familial Dysautonomia, etc)
* significant premorbidity (organ failure, rheumatic disease, etc)
* endotracheal/endobronchial devices including tracheostomy.
* parental refusal to participate in the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
clinical improvement as manifested by resolution of fever and length of hospital admission. | participants will be followed for the duration of hospital stay, an expected average of 10 days

SECONDARY OUTCOMES:
clinical improvement as manifested by respiratory parameters (tachypnea, dyspnea, Fio2),and inflammatory markers. | participants will be followed for the duration of hospital stay, an expected average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: havatzelet yarden-bilavsky, MD, Principal Investigator — schneider children MC of Israel
Locations (1):
- Schneider's medical center of Israel, Petah Tikva, Israel